CLINICAL TRIAL: NCT05604313
Title: Self-reported and Objectively Measured Muscle Tension and Neck Kinematics in Violinists Playing With an Ergonomic and Usual Chinrest: a Randomised Crossover Study
Brief Title: The Effects of Using an Ergonomic Chinrest When Playing the Violin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Axel Muusfeldts fond (Unknown); Region of Southern Denmark (Other); Sygekassernes Helsefond (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 20202000-87
Record Dates: First submitted 2022-10-27; First posted 2022-11-03 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Ergonomics
Keywords: crossover design; neck kinematic; muscle workload; violin playing; performance; comfort

STUDY DESIGN:
Intervention Model Description: We designed a crossover, block randomised (block sizes of 4) and within-subjects experimental design.
Masking Description: This study is open-label, meaning that no masking occurs. The intervention could not be masked (ergonomic equipment testing).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ergonomic chinrest used with low shoulder rest (EC) (Experimental): Participants will play the violin using the ergonomic chinrest with a low Kun Super shoulder rest (EC)
  Interventions: Device: Ergonomic chinrest used with low shoulder rest (EC)
- Do-as-usual (No Intervention): On the test day (crossover study), participants will play with the usual preferred chin and shoulder rest.

INTERVENTIONS:
Device: Ergonomic chinrest used with low shoulder rest (EC) — Participants will play the violin using the ergonomic chinrest with a low Kun Super shoulder rest (EC) for two weeks before the test day (crossover study), measuring upper body kinematic and muscle activity. The novel ergonomic chinrest (Kréddle®, Wyoming, US) is fully adjustable to accommodate each violinist's body type and performance style: regarding height, rotation and tilting. The low Super Kun shoulder rest has been adjusted to be in the lowest position for all legs attached to the violin before the violinists received it. All participants was told not to adjust the shoulder rest but adjust the chinrest.
  Arms: Ergonomic chinrest used with low shoulder rest (EC)

SUMMARY:
A one-day crossover randomised trial was conducted to compare violinists using an ergonomic chinrest (EC) with do-as-usual on muscle activation, kinematics and sound. After two weeks of testing the EC, self-perceived evaluations on comfort, performance, sound, neck alignment and muscle tension were reported in a questionnaire between EC and do-as-usual.

The main question is to answer if:

1. the EC is superior compared to do-as-usual and gives a more aligned neck posture and less muscle tension/dynamic muscle activity
2. the EC is subjectively evaluated as better than do-as-usual regarding self-perceived comfort, performance and sound

DETAILED DESCRIPTION:
The purpose of this study is to investigate the measurement of neck kinematics, muscle activation and sound when using EC and a usual chinrest and, additionally, their self-reported experience of neck alignment, muscle tension, sound experience, performance, and comfort.

It is a crossover, block randomised (block sizes of 4) and within-subjects experimental design performed in one day. The design was made to compare an ergonomic chinrest used with a low shoulder rest (EC) with preferred chin and shoulder rest (do-as-usual) in a randomised order and the effect on muscle activation, kinematics and sound. The study also includes a two-week familiarisation period testing the EC before the test day (crossover design). After these two weeks, a questionnaire was given to register self-reported performance, comfort and sound experience.

Furthermore, the participants were asked in an SMS about what ergonomic equipment they used after half a year (the EC, do-as-usual or other equipment).

On the test day, all participants played with both setup an excerpt of a music piece (second movement from W. A. Mozart's violin concerto no. 5 in A major),

The required sample size was estimated based on a previous feasibility study of either being in an awkward or neutral position with the head. We aimed to recruit 38 professional violinists. A professional violinist was defined as having finished the music conservatory with the violin as the main subject or attending school enrolled in the last years (master/soloist player).

The protocol was initial feasibility tested, and we report this study using the Consolidated Standards of Reporting Trials (CONSORT) 2010 extension to randomised crossover trials.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* speak and write fluently Danish or English
* Professional violinists
* No severe pain symptoms in the neck or upper extremities (<3) scored on a numeric rating scale from 0 (no pain) to 10 (worst perceived pain).

Exclusion Criteria:

* medical conditions that could influence the test result (pacemaker or life-threatening health disorders)
* trauma on the upper cervical spine or upper extremities within the last 12 months
* previous or planned shoulder/neck operation
* severe eczema on the neck and upper extremities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Upper body kinematic was recorded by the device called Vicon | One day
  Neck movement data were collected with Vicon measured in degrees of movement in three anatomical planes: 1) head flexion, 2) head lateral bend, 3) head rotation, 4) trunk flexion, 5) trunk rotation and 6) arm abduction. This measurement was recorded on the test day for both setups while playing a music piece. Furthermore, a test was made on the ROM (head) in a sitting position for all participants before measuring the kinematics during the music piece.
Electromyography was recored with Myon | One day
  Wireless sEMG (Myon 320, AG, Switzerland) was used and placed to measure muscle activity bilaterally from the upper trapezius muscles (UT), upper neck extensor muscles (NE), sternocleidomastoideus muscles (SCM) and on the right medial and left anterior deltoideus muscle (DT). This measurement was recorded on the test day for both setups.
Sound was recorded with Olympus LS-10 stereo digital recorder | One day
  Sound measurement was recorded on the test day for both setups
Self-reported performance score | Two weeks
  Three questions were used for an overall performance score: Have you had difficulty with (within the last 14 days) 1) playing your violin? 2) using your normal technique when playing? 3) playing as well as you would like to? The questions were answered on a 5-point Likert scale from no to impossible. These questions were given after the two-week familiarisation period.
Self-reported comfort score | Two weeks
  Five questions are used for the overall comfort score: How comfortable was (the last 14 days) 1) playing with EC-/ EC+, 2) the height of EC (with your chosen adjustment), 3) the configuration of EC that you have chosen, and 4) the size of the EC chinplate? , 5) the chinrest surface against your skin? The question was answered on a 5-point Likert scale from very comfortable to very uncomfortable. These questions were given after the two-week familiarisation period.
sound quiz | one month
  A quiz with six audio files in a randomised order was sent a month after the test day.
  The quiz was simple: "Do you play using Kréddle (the EC)": yes, no, don't know.
Diary | Two weeks
  Each day during the two-week familiarisation period the violinists had to fill in a diary: written user feedback that will be categorised into positive, negative or neutral feedback. Furthermore about the EC adjustment and their confidence level.
  The adjustment was recorded if they found an adjustment that worked ('Yes', 'No', 'Not yet').
  The confidence level when playing with EC was reported on a 5-point Likert scale (5= very confident, 1=not very confident). 'Very confident' was defined as if the violinist could play the music sheets sent to them also after a break of several days

SECONDARY OUTCOMES:
Adherence | Two weeks
  Adherence to the protocol was recorded from the self-administrated two-week diary.
  Adherence was counted as the number of days playing with the EC out of the two weeks.
Compliance | Two weeks
  Compliance to the protocol was recorded from the self-administrated two-week diary. Compliance for playing with EC was hours played out of total playing time.
Follow-up on which product they are using | 6 month
  After the crossover test day the study ends, but the participants have to answer after a half a year if the are still using EC, do-as-usual or another new setup and if it because they participated in this project. This was answered by a SMS message.
Antroprometrics | One day
  Body measurements were taken on the test day: neck length, arm length, height and shoulder width
Instrument measurement | One day
  On the test day the measurement of the length of the instrument, the shoulder rest height and chin rest height was taken for both setups (EC and do-as-usual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern Denmark, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No